CLINICAL TRIAL: NCT01872338
Title: Mindfulness-Based Cognitive Therapy for Preventing Suicide in Military Veterans
Brief Title: Mindfulness-Based Cognitive Therapy for Suicide Prevention
Acronym: MBCT-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Columbia University (Other); Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 12-134
Record Dates: First submitted 2013-05-10; First posted 2013-06-07 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Suicide
Keywords: suicide prevention; mindfulness-based cognitive therapy; mindfulness meditation; Veterans; safety planning
MeSH Terms: conditions — Suicide; Suicide Prevention | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy + Treatment As Usual (Active Comparator): Psychotherapeutic intervention that integrates mindfulness meditation with Safety Planning, with a specific focus on reducing suicide risk.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy for Suicide
- Treatment As Usual (Other): VA standard care for suicide prevention
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy for Suicide — Psychotherapeutic intervention that integrates mindfulness meditation with Safety Planning, with a specific focus on reducing suicide risk.
  Other Names: MBCT-S
  Arms: Mindfulness-Based Cognitive Therapy + Treatment As Usual
Behavioral: Treatment as usual — VA standard care for suicide prevention
  Arms: Treatment As Usual

SUMMARY:
The purpose of this study is to test a psychotherapeutic intervention that integrates cognitive therapy and mindfulness meditation techniques to prevent suicide in military Veterans.

DETAILED DESCRIPTION:
Every month the VA becomes aware of approximately 1,100 Veterans in VA care who attempt suicide. While the VA has implemented a comprehensive, multifaceted suicide prevention approach, it has yet to implement nationally any evidence-based psychotherapies targeting suicide, a gap due largely to the dearth of evidence-based therapies for suicide. Primary aims of this proposal are to conduct a randomized controlled trial testing an adaptation of a cognitive-behavioral intervention, Mindfulness-Based Cognitive Therapy (MBCT), for Veterans on the VA's High Risk for Suicide List. The investigators' adapted version of MBCT for suicide (MBCT-S) integrates mindfulness meditation techniques with the VA Safety Plan to enhance patients' awareness of suicide triggers and appropriate coping strategies. This study has the potential to increase the range of cost effective treatment alternatives for the large number of suicidal Veterans for whom evidence-based therapies are severely limited.

ELIGIBILITY:
Inclusion Criteria:

The following criteria were formulated to recruit a sample at high risk for suicide behavior.

* The subject has experienced a suicidal event during the past 30 days. A suicidal event involves

  * 1) psychiatric hospitalization due to suicidal risk,
  * 2) psychiatric hospitalization if subject was already on the High Risk for Suicide List,
  * 3) suicidal ideation with suicidal intent,
  * 4) suicidal preparatory behaviors, or
  * 5) actual, interrupted, or aborted suicide attempt.

AND

* The subject is on or will be placed on the VA High Risk for Suicide List

  * OR The subject had an actual, interrupted, or aborted attempt in the last year
  * OR In the study clinician's opinion (i.e., Masters or Doctoral level study personnel with formal mental health training) in consultation with the PI, the suicidal event is significant enough to warrant treatment to reduce suicidal risk.

Exclusion Criteria:

* cognitive deficits that decrease the likelihood of benefit from MBCT-S
* severe symptoms of hallucinations or delusions
* disorganized or disruptive behaviors
* medically unstable
* current mindfulness-based psychotherapy or receipt of 2 or more sessions of a mindfulness-based psychotherapy in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Interian, PhD, Principal Investigator — Lyons Campus of the VA New Jersey Health Care System, Lyons, NJ
Locations (2):
- United States (2):
  - East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey
  - Lyons Campus of the VA New Jersey Health Care System, Lyons, NJ, Lyons, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Interian A, Miller R, Dave C, Latorre M, St Hill L, King A, Boschulte DR, Kline A, Siegel D, Sedita MM, Chesin MS. Examining the Occurrence and Clinical Impact of Difficult Experiences that Emerge during a Mindfulness-Based Intervention among Individuals at High-Risk of Suicide. Mindfulness (N Y). 2024 Jun 18;15:1701-1712. PMID 40134457
- [Derived] Interian A, Chesin MS, Stanley B, Latorre M, St Hill LM, Miller RB, King AR, Boschulte DR, Rodriguez KM, Kline A. Mindfulness-Based Cognitive Therapy for Preventing Suicide in Military Veterans: A Randomized Clinical Trial. J Clin Psychiatry. 2021 Aug 31;82(5):20m13791. doi: 10.4088/JCP.20m13791. PMID 34464524

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-Based Cognitive Therapy + Treatment As Usual | Treatment As Usual
Started | 66 | 69
Completed | 46 | 69
Not Completed | 20 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Cognitive Therapy + Treatment As Usual | Treatment As Usual | Total
Number analyzed (Participants) | 66 | 69 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.54 (13.2) | 45.97 (14.3) | 46.96 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 59 | 60 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  RACE/ETHNICITY: White | 30 | 31 | 61
  RACE/ETHNICITY: Black | 15 | 21 | 36
  RACE/ETHNICITY: Asian, American Indian, or other | 7 | 2 | 9
  RACE/ETHNICITY: Latino | 14 | 15 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 69 | 135
Suicide Attempt History [Count of Participants; unit: Participants]
  none | 9 | 12 | 21
  one | 21 | 17 | 38
  multiple | 36 | 40 | 76

OUTCOME MEASURES:

1. Primary Outcome: Suicide Event
Description: The investigators define "event" broadly as a range of suicidal behaviors defined according to the VA's Self-Directed Violence Classification System (SDVCS). Based on the SDVCS, an event may include self-directed violence, with or without injury, in which evidence of suicidal intent is clear or undetermined; or suicidal preparatory behaviors. The study definition of a suicide event also includes suicidal ideation resulting in the need for emergency care or psychiatric hospitalization.
Time Frame: 12-months post-baseline
Population: Total number of suicidal events within the 12-month observation period by study condition.
Measure: Number; unit: count of events
Arm/Group | Mindfulness-Based Cognitive Therapy + Treatment As Usual | Treatment As Usual
Number analyzed (Participants) | 66 | 69
count of events | 44 | 92
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy + Treatment As Usual vs Treatment As Usual; Test type: Superiority; p = .015, negative binomial regression; Incident Rate Ratio = .50, 95% CI 2-sided [.29 to .87]

2. Secondary Outcome: Suicide Attempt
Description: Defined as deliberate self-directed violence with injury or potential for injury and with explicit/implicit suicidal intent
Time Frame: 12 months post-baseline
Population: count of suicide attempts over 12-month period by study condition
Measure: Number; unit: count of suicide attempts
Arm/Group | Mindfulness-Based Cognitive Therapy + Treatment As Usual | Treatment As Usual
Number analyzed (Participants) | 66 | 69
count of suicide attempts | 11 | 27
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy + Treatment As Usual vs Treatment As Usual; Test type: Superiority; p = .01, negative binomial regression; Incident Rate Ratio = .43, 95% CI 2-sided [.22 to .82]

3. Secondary Outcome: Suicidal Ideation
Description: clinician-administered Scale for Suicide Ideation (SSI), 0-38, higher score = higher suicidal ideation.
Time Frame: Baseline, 4 weeks (mid-treatment), 8 weeks (treatment-completion), 6 months and 12-months post-baseline
Population: Linear mixed models, examining change from baseline over 12 months (5 assessments total), with effect of interest being time*cond interaction.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy + Treatment As Usual | Treatment As Usual
Number analyzed (Participants) | 66 | 69
score on a scale
  Time 1 | 12.4 (1.2) | 11.2 (1.2)
  Time 2 | 5.8 (1.2) | 6.1 (1.2)
  Time 3 | 4.8 (1.1) | 4.7 (1.0)
  Time 4 | 6.1 (1.1) | 3.3 (1.0)
  Time 5 | 3.8 (.9) | 2.3 (.8)
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy + Treatment As Usual vs Treatment As Usual; Test type: Superiority; p = .34, Regression, Linear; repeated measures, overall time by condition effect

4. Secondary Outcome: Hopelessness
Description: Hopelessness will be measured using the Beck Hopelessness Scale, score range 0-20, with higher scores indicating more hopelessness.
Time Frame: Baseline, 4 weeks (mid-treatment), 8 weeks (treatment-completion), 6 months and 12-months post-baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy + Treatment As Usual | Treatment As Usual
Number analyzed (Participants) | 66 | 69
score on a scale
  Time 1 | 13.4 (.7) | 11.8 (.7)
  Time 2 | 8.4 (.9) | 8.1 (.8)
  Time 3 | 7.4 (.9) | 8.3 (.9)
  Time 4 | 8.0 (.9) | 7.7 (.9)
  Time 5 | 8.7 (1.0) | 8.6 (.9)
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy + Treatment As Usual vs Treatment As Usual; Test type: Superiority; p = .23, Regression, Linear — repeated measures, overall time by condition effect

ADVERSE EVENTS:
Time Frame: 12-month study participation period
Description: all serious adverse events were reported to IRB and reviewed by a DSMB
Arm/Group | Mindfulness-Based Cognitive Therapy + Treatment As Usual | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 3/66 | 1/69
Serious Adverse Events (participants affected / at risk) | 31/66 | 40/69
Other Adverse Events (participants affected / at risk) | 4/66 | 4/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness-Based Cognitive Therapy + Treatment As Usual (N=66) | Treatment As Usual (N=69)
Psychatric Adverse Events (Psychiatric disorders) | 26 (45) | 37 (85)
Medical SAE (Cardiac disorders) | 3 (5) | 3 (3) — **no adverse events were determined by IRB to be related to the research procedures or intervention
Medical SAE (Endocrine disorders) | 2 (2) | 0 (0) — **no adverse events were determined by IRB to be related to the research procedures or intervention
Medical SAE (Gastrointestinal disorders) | 2 (2) | 1 (1) — **no adverse events were determined by IRB to be related to the research procedures or intervention
Medical SAE (General disorders) | 1 (1) | 1 (1) — **no adverse events were determined by IRB to be related to the research procedures or intervention
Medical SAE (Infections and infestations) | 0 (0) | 1 (1) — **no adverse events were determined by IRB to be related to the research procedures or intervention
Medical SAE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — **no adverse events were determined by IRB to be related to the research procedures or intervention
Medical SAE (Nervous system disorders) | 2 (2) | 1 (1) — **no adverse events were determined by IRB to be related to the research procedures or intervention
Medical SAE (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) — **no adverse events were determined by IRB to be related to the research procedures or intervention
Medical SAE (Surgical and medical procedures) | 3 (3) | 0 (0) — **no adverse events were determined by IRB to be related to the research procedures or intervention
Medical SAE (Vascular disorders) | 0 (0) | 1 (1) — **no adverse events were determined by IRB to be related to the research procedures or intervention
SAE Other (Social circumstances) | 1 (1) | 2 (2) — **no adverse events were determined by IRB to be related to the research**
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness-Based Cognitive Therapy + Treatment As Usual (N=66) | Treatment As Usual (N=69)
Psychiatric other (not including serious) (Psychiatric disorders) | 4 (6) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT01872338/Prot_SAP_000.pdf